CLINICAL TRIAL: NCT02534688
Title: Effectiveness of Levonorgestrel-intrauterine System (LNG-IUS) Versus Depot Medroxyprogesterone Acetate (DMPA) in Treatment of Pelvic Pain in Clinically Diagnosed Endometriotic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kamolrat Daoudom, Effectiveness of levonorgestrel-intrauterine system (LNG-IUS) versus depot medroxyprogesterone acetate (DMPA) in treatment of pelvic pain in clinically diagnosed endometriotic patients, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kingchulalongkorn
Record Dates: First submitted 2015-08-19; First posted 2015-08-28 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — N,N-dimethyl-4-anisidine

ARMS (2):
- LNG-IUS group (Experimental): Single intervention LNG IUS
  Interventions: Drug: LNG-IUS
- DMPA group (Experimental): Three intervention DmPA 12 wk apart
  Interventions: Drug: DMPA

INTERVENTIONS:
Drug: LNG-IUS
  Arms: LNG-IUS group
Drug: DMPA
  Arms: DMPA group

SUMMARY:
randomized controlled trial

Eligiblility criteria Provisional diagnosis Clinical presentation Progressive dysmenorrhea Chronic pelvic pain Deep dyspareunia Evidences of endometriosis Endometriotic nodule Cul-de-sac nodularity Endometrioma detected by ultrasonography size < 4 cm

Inclusion criteria Female age 18-45 yr Moderate to severe pelvic pain categorized by VAS >50 Previous sexual intercourse

Exclusion criteria Co-existing other genital tract disease associated pain Previous hormonal use within 3 months History of DMPA treatment failure WHO eligibility criteria 2009 for DMPA and LNG-IUS Category 3,4 Fertility desire in upcoming 1 year

Primary objective To compare efficacy of pain control in endometriosis associated pelvic pain between LNG-IUS and DMPA

Secondary objective To compare side effect, continuation rate, satisfaction and quality of life between LNG-IUS and DMPA in treatment of endometriosis associated pelvic pain

Primary outcome Severity of pelvic pain Measured by VAS score 0 mean no pain 100 mean most pain

Secondary outcomes Vaginal bleeding pattern Side effects of systemic progestogen Lipid profiles Weight gain Quality of life Measured by quesionaire SF36 Satisfaction Measrured by linket scale 0-4 0 mean very dissatisfied 1 dissatisfied 2 not satisfied and dissatiffied 3 satisfied 4 very satisfied Continuation rate Endometrioma size reduction

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-45 yr
* Moderate to severe pelvic pain categorized by VAS >50
* Previous sexual intercourse

Exclusion Criteria:

* Co-existing other genital tract disease associated pain
* Previous hormonal use within 3 months
* History of DMPA treatment failure
* WHO eligibility criteria 2009 for DMPA and LNG-IUS Category 3,4
* Fertility desire in upcoming 1 year

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Severity of pelvic pain : measured by visual analog scale | 6 months

SECONDARY OUTCOMES:
Quality of life measured by Quesionaire SF 36 Thai version | 6 months
Lipid profile : total cholesterol, triglyceride, LDL, HDL | 6months
  Measured by blood collection in mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memmorial hospital, Bangkok, Bangkok, Thailand